CLINICAL TRIAL: NCT00866775
Title: Double-Blind, Randomized, Historical Control Study of the Safety and Efficacy of Eslicarbazepine Acetate Monotherapy in Subjects With Partial Epilepsy Not Well Controlled by Current Antiepileptic Drugs
Brief Title: Safety and Efficacy of Eslicarbazepine Acetate Monotherapy in Subjects With Partial Epilepsy Not Well Controlled by Current Antiepileptic Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 093-045
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Epilepsy With Simple or Complex Partial Onset Seizures
Keywords: Seizure; Epilepsy; Anticonvulsant; Historical Control; Monotherapy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eslicarbazepine 1600 mg QD (Experimental): Subjects randomized to 1600 mg QD of eslicarbazepine acetate will titrate from 600 mg QD (Day 0) to 1200 mg QD (Week 1) to 1600 mg QD (Weeks 2-18)
  Subjects may continue in an open-label extension study with a starting dose of 1600 mg QD, or taper off study drug at the completion of this study The treatment period for subjects entering the open label extension study is up to 9 study visits over 18 weeks. The treatment period for subjects not entering the open-label extension study is up to 10 study visits over 19 weeks.
  Interventions: Drug: Eslicarbazepine acetate
- Eslicarbazepine 1200 mg QD (Experimental): Subjects randomized to 1200 mg QD eslicarbazepine acetate will titrate from 400 mg QD (Day 0) to 800 mg QD (week 1) to 1200 mg QD (weeks 2-18)
  Subjects may continue in an open-label extension study with a starting dose of 1600 mg QD, or taper off study drug at the completion of this study The treatment period for subjects entering the open label extension study is up to 9 study visits over 18 weeks. The treatment period for subjects not entering the open-label extension study is up to 10 study visits over 19 weeks.
  Interventions: Drug: Eslicarbazepine acetate

INTERVENTIONS:
Drug: Eslicarbazepine acetate — 1600 mg QD
  Arms: Eslicarbazepine 1600 mg QD
Drug: Eslicarbazepine acetate — 1200 mg QD
  Arms: Eslicarbazepine 1200 mg QD

SUMMARY:
This is an 18-week, double-blind, multicenter study with gradual conversion from previous antiepileptic therapy to eslicarbazepine acetate monotherapy in subjects with partial epilepsy.

DETAILED DESCRIPTION:
This is an 18-week, double-blind, randomized, historical control, multicenter study with gradual conversion to monotherapy in subjects with partial onset seizures who are not well controlled by current AEDs. The 18 week double-blind treatment period consists of a 2-week period for titration of study drug, 6-week period for taper or conversion off AEDs, and a 10-week monotherapy period. Subjects not entering an optional open-label extension study will enter a 1-week period to taper off study drug followed by an end of study visit (week 19). This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of partial epilepsy as defined in the Classification of Seizures of the International League Against Epilepsy (ILAE) (simple partial seizures with observable motor component, or complex, with or without secondary generalization) a. Medical history of seizures; b. Absence of confounding factors (pseudoseizures, syncope); c. Documented EEG recording (done within 5 years prior to screening) consistent with focal onset epilepsy.
* Documented CT or MRI scan conducted within 10 years prior to screening, showing the absence of a progressive structural abnormality (eg, tumor). Mesial temporal sclerosis is acceptable.
* ≥4 partial onset seizures during the 8 weeks prior screening with no 28-day seizure free period.
* Stable treatment with 1-2 AEDs during the last 4 weeks prior to screening.
* Subjects must have the ability to comprehend the informed consent form and be willing to provide informed consent. For subjects who are unable to comprehend the written consent, a witness/caregiver who is able to describe and provide an understanding of the informed consent to the subject must sign the consent form on behalf of the subject.
* Subjects must give written informed consent prior to participation in the study. For subjects <18 years of age, the informed consent must be signed by the subject's parent or legal guardian, and, when appropriate and/or required by state or local law, minor subjects must give written informed assent prior to participation in the study. Subjects of Asian ancestry are required to give written informed consent for genotyping. All subjects must sign a HIPAA Form. All females of child bearing potential must also sign the "Women of Childbearing Potential" Addendum.
* A female subject is eligible to enter and participate in the study if she is of: a. Non-childbearing potential (ie, physiologically incapable of becoming pregnant, including any female who is pre-menarchal or post-menopausal); b. Child-bearing potential (all females ≤65 years of age), has a negative pregnancy test at screening and agrees to satisfy contraception requirements.

Exclusion Criteria:

* Subjects with only simple partial seizures without a motor component.
* Presence of generalized seizure syndromes (eg, juvenile myoclonic epilepsy or Lennox-Gastaut syndrome).
* History of pseudo-seizures.
* Current seizures related to an acute medical illness.
* Seizures secondary to metabolic, toxic or infectious disorder or drug abuse.
* Status epilepticus within 2 years prior to screening.
* Seizures only occurring in a cluster pattern.
* Subjects taking 2 of the following sodium channel blocking AEDs: phenytoin, carbamazepine, oxcarbazepine, or lamotrigine.
* Subjects taking 2 AEDs with both being in the upper dose range (defined as approximately two-thirds of the defined daily dose).
* Subjects taking more than 2 AEDs.
* Subjects with progressive structural central nervous system lesion or progressive encephalopathy.
* Psychiatric exclusion criteria: subjects with history of suicide attempt in last 2 years; major depressive episode within last 6 months; abuse of alcohol or substance abuse in last 2 years; significant psychiatric disorder or recurrent episodes of severe depression within 2 years prior to screening.
* Medical exclusion criteria: known renal insufficiency or subject with estimated creatinine clearance [CrCL] <60 mL/min based on serum creatinine using the Cockcroft-Gault formula.
* Clinical and laboratory exclusion criteria: Subjects of Asian ancestry who tests positive for the presence of the HLA-B*1502 allele.
* Subjects who have been on benzodiazepines, phenobarbital, or primidone on a regular basis within 3 months prior to screening.
* Subjects taking antipsychotics, tricyclic antidepressants, anxiolytics, sedative hypnotics including non-benzodiazepines, central opioid agonists/antagonists, monoamine oxidase inhibitors (MAOIs) within at least 5 half lives (or for at least 2 weeks whichever is longer) prior to randomization.
* Subjects presently on felbamate or vigabatrin
* Female subjects who are currently breastfeeding or intending to breastfeed during study period.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (106):
- United States (103):
  - Norwood Neurology, Birmingham, Alabama
  - Greystone Neurology Center, Birmingham, Alabama
  - USA Neurology, Mobile, Alabama
  - Neurology Clinic, P.C., Northport, Alabama
  - Clinical Research Consortium, Phoenix, Arizona
  - Clinical Research Consortium - Arizona, Phoenix, Arizona
  - Xenoscience Inc., Phoenix, Arizona
  - Arizona Neurological Institute, Sun City, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - K & S Professional Research Services, Little Rock, Arkansas
  - Sutter East Bay Medical Foundation, Berkley, California
  - Synergy Escondido, Escondido, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - Faculty of Physicians & Surgeons of Loma Linda University, Loma Linda, California
  - Loma Linda University, Loma Linda, California
  - American Institute of Research, Los Gatos, California
  - Northridge Neurological Center, Northridge, California
  - Yafa Minazad, DO, Pasadena, California
  - Neurological Research Institute, Santa Monica, California
  - American Institute of Research, Whittier, California
  - Anschutz Outpatient Pavilion, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Associated Neurologists, PC, Danbury, Connecticut
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Miami Clinical Research, Coral Gables, Florida
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Infiniti Clinical Research, LLC, Hollywood, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - Neurology Associates, PA, Maitland, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - San Marcus Research Clinic, Miami, Florida
  - Neurosciences Consultants, LLC, Miami, Florida
  - Neurological Services Orlando, Orlando, Florida
  - Pediatric Neurolog, PA, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Pediatric Epilepsy & Neurology Specialists, PA, Tampa, Florida
  - Florida Comprehensive Epilepsy and Seizure Disorder Center, Tampa, Florida
  - Vero Neurology, Vero Beach, Florida
  - Palm Beach Clinical Research Network LLC, Wellington, Florida
  - Peachtree Neurological Clinic, Atlanta, Georgia
  - Emory University Department of Neurology, Atlanta, Georgia
  - PANDA Neurology and Atlanta Headache Specialists, Atlanta, Georgia
  - Harbin Clinic, Rome, Georgia
  - GA Neurology and Sleep Medicine Associates, Suwanee, Georgia
  - Consultants in Epilepsy and Neurology, PLLC., Boise, Idaho
  - Rush University, Chicago, Illinois
  - UCMC, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - McFarland Clinic, PC, Ames, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Epilepsy Research LLC, Lexington, Kentucky
  - North Oaks Neurology, Hammond, Louisiana
  - MMP Neurology, Scarborough, Maine
  - John Hopkins University, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Massachusetts General Hospital Epilepsy Service - WACC, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - The Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Cooper University Health System, Camden, New Jersey
  - Cooper University Health System, Cherry Hill, New Jersey
  - NJ Neuroscience Center, Edison, New Jersey
  - Institute of Neurology and Neurosurgery at St. Bamabas, Suite 101, Livingston, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - Winthrop University Hospital, Mineola, New York
  - Beth Israel Medical Center, New York, New York
  - Clinilabs Inc., New York, New York
  - University of Rochester, Rochester, New York
  - The Neurology Institute, Charlotte, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Wake Forest University, Winstom-Salem, North Carolina
  - Northern Ohio Neurosciences, Bellevue, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - 5929 N. May Ave., Oklahoma City, Oklahoma
  - Providence Medical Group, Medford, Oregon
  - Children's Hospital Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburg of UPMC, Pittsburgh, Pennsylvania
  - Gus Stratton / Neurology, Cranston, Rhode Island
  - Mid-South Physcians Group, Germantown, Tennessee
  - Access Clinical Trials, Nashville, Tennessee
  - VU Department of Neurology, Nashville, Tennessee
  - Neurology Associates of Arlington, PA, Arlington, Texas
  - Texas Neurology, PA, Dallas, Texas
  - Neurological Clinic of Texas P.A., Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - UT Health Science Center at Houston, Houston, Texas
  - Todd Swick, MD, PA, Houston, Texas
  - Neurology Associates of Arlington, PA, Mansfield, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Sentara Neurology Specialists, Norfolk, Virginia
  - Neurological Associates of Washington/Clinical Trials of America Inc., Bellevue, Washington
  - Rainier Clinical Research Center, Inc., Renton, Washington
  - Pacific Medical Centers, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (3):
  - London Health Sciences Center, London, Ontario
  - Neuro-Epilepsy Clinic, Greenfield Park, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Background] Sperling MR, Harvey J, Grinnell T, Cheng H, Blum D; 045 Study Team. Efficacy and safety of conversion to monotherapy with eslicarbazepine acetate in adults with uncontrolled partial-onset seizures: a randomized historical-control phase III study based in North America. Epilepsia. 2015 Apr;56(4):546-55. doi: 10.1111/epi.12934. Epub 2015 Feb 16. PMID 25689448

RESULTS

PARTICIPANT FLOW:
Groups:
- Eslicarbazepine 1200 mg QD: Subjects randomized to 1200 mg QD eslicarbazepine will titrate from 400 mg (Week 1) to 800 mg (Week 2) to 1200 mg (Weeks 3-18) QD and taper down from 1200 mg to 600 mg QD 3 days after the end of Week 18.
  .
- Eslicarbazepine 1600 mg QD: Subjects randomized to 1600 mg QD of eslicarbazepine will titrate from 600 mg (Week 1) to 1200 mg (Week 2) to 1600 mg (Weeks 3-18) QD and taper down from 1600 mg to 800 mg QD 3 days after the end of Week 18.
Period: Overall Study
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Started | 65 | 128
Completed | 29 | 76
Not Completed | 36 | 52
Not completed — Adverse Event | 5 | 19
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 4
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawal by Subject | 4 | 4
Not completed — met exit criteria | 23 | 17
Not completed — discontinued due to communication error | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD | Total
Number analyzed (Participants) | 65 | 128 | 193
Age, Customized [Number; unit: participants]
  less than 18 years | 4 | 2 | 6
  18-39 years | 31 | 61 | 92
  40-65 years | 29 | 61 | 90
  greater than 65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 67 | 101
  Male | 31 | 61 | 92
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alsaka Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 18 | 22
  White | 53 | 94 | 147
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 5 | 6
  United States | 64 | 123 | 187

OUTCOME MEASURES:

1. Primary Outcome: Cumulative 112-day Exit Rate as Estimated by Kaplan-Meier Method
Description: Cumulative exit rate was defined as the proportion of subjects meeting at least one of the five exit criteria over a 16-wk study period (start of Antiepilectic Drugs(AED) taper/conv.period (Wk 3 to end of double blind monotherapy period (Wk 18)):1.One episode of status epilepticus.2.One secondary general partial seizure (in subjects who did not have gen. seizures during 6 months prior to screening).3.A two fold increase in any consecutive 28 day seizure rate compared to the highest consecutive 28 day seizure rate during the 8 wk baseline period. 4.A two fold increase in any consecutive 2 day seizure rate compared to the highest consecutive 2 day seizure rate during the 8 wk baseline period. If the highest number of seizures in any consecutive 2 day period during the 8 wk baseline was 1 then 3 seizures in a consecutive 2 day period was required to exit.5.Worsening of seizures or increase in seizure frequency considered serious or requiring intervention as judged by the Investigator.
Time Frame: Week 3 to Week 18
Population: efficacy population
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
proportion of participants | 0.444 [0.3252 to 0.5832] | 0.287 [0.2124 to 0.3813]

2. Secondary Outcome: Percentage of Subjects That Are Seizure-free During the 10-week Double-blind Monotherapy Treatment Period.
Description: Seizure-free subjects during the monotherapy period were determined as subjects who had seizure assessments during the monotherapy period, and did not have any seizures in the 10 weeks between Visits 6 and 9 (Weeks 9 through 18). Subjects who discontinued during this period were considered not seizure-free even if they were seizure-free at the time of discontinuation, i.e., to be considered seizure-free, subjects must complete the 10-week period without any seizures.
Time Frame: Weeks 9 through 18
Population: efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
percentage of participants | 8.3 [2.8 to 18.4] | 7.6 [3.5 to 14.0]

3. Secondary Outcome: Percentage of Subjects Seizure-free During the Last 4 Weeks on Eslicarbazepine Acetate Monotherapy.
Description: Seizure-free subjects during the last four weeks of monotherapy were determined as subjects who had seizure assessments during the 4 weeks between Visits 8 and 9 (Weeks 15 through 18), and did not have any seizures.
Time Frame: Weeks 15 through 18
Population: efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
percentage of participants | 13.3 [5.9 to 24.6] | 14.4 [8.6 to 22.1]

4. Secondary Outcome: Completion Rate
Description: Subjects completing the study were determined as subjects who completed the 18 weeks of double-blind treatment.
Time Frame: Week 1 to Week 18
Population: efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
percentage of participants | 48.3 [35.2 to 61.6] | 64.4 [55.1 to 73.0]

5. Secondary Outcome: Completion Rate During the 10 Weeks of Monotherapy
Description: Monotherapy completion rate was defined as the proportion (%) of subjects entering the monotherapy period who completed the 10 weeks of monotherapy treatment.
Time Frame: Weeks 8 through 18
Population: efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 45 | 93
percentage of participants | 64.4 [48.8 to 78.1] | 81.7 [72.4 to 89.0]

6. Secondary Outcome: Time on Eslicarbazepine Acetate Monotherapy.
Description: The start of the monotherapy period was defined as the date of termination of all other AEDs while taking study monotherapy medication. Time on monotherapy was defined from the start of monotherapy period to the last dose of monotherapy treatment.
Time Frame: Week 8 to Week 18
Population: efficacy population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
days | NA [NA to NA] — median not calculable due to lack of events | NA [NA to NA] — median not calculable due to lack of events

7. Secondary Outcome: Change in Seizure Frequency From Baseline.
Description: The relative (%) change in standardized seizure frequency was evaluated for four periods: titration (Weeks 1 to 2), AED taper/conversion (Weeks 3 to 8), monotherapy (Weeks 9 to 18), and double-blind (Weeks 1 to 18).
Time Frame: Week 0 to Week 18, Double-blind: weeks 1to 18; baseline:weeks-8 to -1; Titration: weeks 1 to 2; AED taper/conversion:weeks 3 to 8; monotherapy: weeks 9 to 18
Population: efficacy population (ESL 1200 mg) Double-blind: 60;Titration: 60; AED taper/conversion: 60; Monotherapy: 43 (ESL 1600 mg) Double-blind: 118; Titration: 118; AED taper/conversion:114; Monotherapy:93
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
percent change
  Relative (%) change from baselne for DB period | -30.9 [-63.3 to 30.9] | -41.5 [-65.6 to -9.5]
  Relative (%) change from baseline -tiration period | -29.6 [-100.0 to 1.8] | -52.4 [-100.0 to -11.4]
  Relative (%) change from baseline -AED t/c period | -30.2 [-69.5 to 25.9] | -39.7 [-78.3 to 1.6]
  Relative (%) change from baseline - mono period | -48.7 [-73.2 to 43.3] | -38.6 [-77.1 to -7.9]

8. Secondary Outcome: Responder Rate (Proportion [%] of Subjects With a ≥50% Reduction of Seizure Frequency From Baseline).
Description: Responder rate was defined as the proportion (%) of subjects with a ≥ 50% reduction of seizure frequency from baseline. This analysis was done for the titration (Weeks 1 to 2), AED taper/conversion (Weeks 3 to 8), monotherapy (Weeks 9 to 18), and double-blind (Weeks 1 to 18) periods.
Time Frame: Week 0 to Week 18, Double blind: weeks to 8; baseline:weeks -8 to -1; titration: weeks 1 to 2; AED taper/conversion: weeks 3 to 8; monotherapy: weeks 9 to 18
Population: efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
percentage of participants
  Responder rate during double blind period | 36.7 [24.6 to 50.1] | 39.8 [30.9 to 49.3]
  Responder rate during the titration period | 46.7 [33.7 to 60.0] | 51.7 [42.3 to 61.0]
  Responder Rate during the AED T/C period | 41.7 [29.1 to 55.1] | 43.2 [34.1 to 52.7]
  Responder rate during monotherapy period | 35.0 [23.1 to 48.4] | 32.2 [23.9 to 41.4]

9. Secondary Outcome: Percentage of Subjects Reaching Each of the Exit Events.
Description: The percentage of subjects reaching each of the 5 exit criteria. 1.One episode of status epilepticus.2.One secondary general partial seizure (in subjects who did not have gen. seizures during 6 months prior to screening).3.A two fold increase in any consecutive 28 day seizure rate compared to the highest consecutive 28 day seizure rate during the 8 wk baseline period. 4.A two fold increase in any consecutive 2 day seizure rate compared to the highest consecutive 2 day seizure rate during the 8 wk baseline period. If the highest number of seizures in any consecutive 2 day period during the 8 wk baseline was 1 then 3 seizures in a consecutive 2 day period was required to exit.5.Worsening of seizures or increase in seizure frequency considered serious or requiring intervention as judged by the Investigator.
Time Frame: Week 1 to Week 18
Population: efficacy population
Measure: Number; unit: percentage of participants
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
percentage of participants
  exit criterion 1 | 0 | 0.8
  exit criterion 2 | 6.7 | 0.8
  exit criterion 3 (investigator prog. assessment) | 10.0 | 4.2
  exit criterion 3 (sponsors prog. assessment) | 8.3 | 5.9
  exit criterion 4 (investigaor prog. assessment) | 8.3 | 5.1
  exit criterion 4 (sponsor prog. assessment) | 10.0 | 5.9
  exit criterion 5 | 13.3 | 3.4

10. Secondary Outcome: Change in Total Score From Baseline in 31-Item Quality of Life in Epilepsy (QOLIE-31).
Description: The QOLIE-31 overall score was obtained by using a weighted average of multi-item scale scores. The recorded responses were converted to 0-100 point scales. The mean of the individual item scores in each subgroup were calculated, with higher converted scores reflecting better quality of life.
Time Frame: Week 0 to Week 18, baseline: day 0: End of AED taper/conversion period: end of week 8; End of monotherapy period: end of week 18
Population: the numbers analyzed represent all participants for whom data were available at baseline (ESL 1200 mg)Change from baseline to end of AED taper/conversion period: 39;Change from baseline to end of monotherapy period:36 (ESL1600 mg) Change from baseline to end of AED taper/conversion period: 86;Change from baseline to end of monotherapy period: 86
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 54 | 113
units on a scale
  Change from baseline to end of AED T/C pd n=39,86 | 3.2 (10.75) | 6.3 (12.42)
  change from baseline to end of mono. pd n=36,86 | 7.8 (13.78) | 6.4 (12.64)

11. Secondary Outcome: Change in Total Score From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS).
Description: The total score of MADRS is defined as the sum of all individual symptom scores, ranging from 0 to 60, higher score indicates more severe depression. Each of the 10 symptoms of depression on MADRS was measured on a scale of 0 to 6 with 0 representing the lowest severity of the symptom and 6 representing the highest severity
Time Frame: Week 0 to Week 18; Baseline: day 0; End of AED taper/conversion period: end of week 8; End of monotherapy period: end of week 18
Population: efficacy population (ESL 1200 mg) Change from baseline to end of AED taper/conversion period: 45; Change from baseline to end of monotherapy period: 41 (ESL 1600 mg) Change from baseline to end of AED taper/conversion period: 92; Change from baseline to end of monotherapy period: 91
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 60 | 118
units on a scale
  Change from baseline to AED T/C period | -0.4 (4.35) | -2.0 (5.99)
  Change from baseline to end of mono period | -1.1 (5.55) | -2.4 (5.77)

12. Secondary Outcome: Change in Total Score From Baseline in MADRS in Those Subjects With a MADRS Score of ≥14 at Randomization.
Description: as for outcome 11
Time Frame: Week 0 to Week 18, Baseline: Day 0; End of AED taper/conversion period: end of week 8; End of monotherapy period: end of week 18
Population: efficacy population (ESL 1200 mg) Change from baseline to end of AED taper/conversation period: 7; Change from baseline to end of monotherapy period: 6 (ESL 1600 mg) Change from baseline to end of AED taper/conversation period: 13; Change from baseline to end of monotherapy period: 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 9 | 17
units on a scale
  Change from baseline to AED T/C pd n=7,13 | -1.3 (3.86) | -7.9 (9.81)
  Change from baseline to end of mono pd n=6,13 | -6.8 (6.71) | -9.6 (8.72)

13. Secondary Outcome: Percentage of Subjects With Increase of Body Weight >= 7%
Time Frame: 18 Week Double-blind treatment period
Population: ITT population
Measure: Number; unit: Percentage of participants
Groups:
- Eslicarbazepine 1200 mg QD: Subjects randomized to 1200 mg QD eslicarbazepine acetate will titrate from 400 mg (Week 1) to 800 mg (Week 2) to 1200 mg (Weeks 3-18) QD and taper down from 1200 mg to 600 mg QD 3 days after the end of Week 18.
  .
- Eslicarbazepine 1600 mg QD: Subjects randomized to 1600 mg QD of eslicarbazepine acetate will titrate from 600 mg (Week 1) to 1200 mg (Week 2) to 1600 mg (Weeks 3-18) QD and taper down from 1600 mg to 800 mg QD 3 days after the end of Week 18.
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 65 | 128
Percentage of participants | 2 | 9

14. Secondary Outcome: Proportion (%) of Subjects With Normal Baseline Sodium Reaching Blood Sodium ≤135 mmol/L, ≤130 mmol/L, and ≤125 mmol/L
Description: Proportion (%) of Subjects With Normal Baseline Sodium Reaching Blood Sodium ≤135 mmol/L, ≤130 mmol/L, and ≤125 mmol/L
Time Frame: 18 Week Double-blind treatment period
Population: ITT population
Measure: Number; unit: Percent
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 65 | 128
Percent
  ≤ 135 and > 130 mEq/L | 29 | 61
  ≤ 13- amd > 125 mEq/L | 6 | 11
  ≤125 mEq/L | 3 | 5

15. Secondary Outcome: Proportion (%) of Events in Each Classification of the Columbia Suicide Severity Rating Scale (C SSRS).
Time Frame: 18 Week Double-blind treatment period
Population: ITT population
Measure: Number; unit: Percent of participants
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 65 | 128
Percent of participants
  Actual Attempt | 0 | 0
  Non-suicidal Self-Injurious Behavior | 0 | 0
  Interrupted Attempt | 1.5 | 0
  Aborted Attempt | 0 | 0
  Preparatory Attempts | 1.5 | 0
  SuicidalBehavior | 0 | 0
  Wish to be Dead | 4.6 | 3.1
  Non-specific Active Suicidal Thoughts | 4.6 | 0.8
  Act. Suicidal Idea. w/any method-no intent to act | 1.5 | 0.8
  Act. Suicidal Idea.w/any method-some intent to act | 0 | 0
  Act. Suicidal Idea. w/any method-Spec. Plan to act | 0 | 0

16. Secondary Outcome: Standardized Seizure Frequency (SSF) by Period
Description: Seizure frequency was evaluated by using a standardized frequency per 4 weeks (28 days). It was evaluated for five periods: baseline (Weeks -8 to -1), titration (Weeks 1 to 2), AED taper/conversion (Weeks 3 to 8), monotherapy (Weeks 9 to 18), and double-blind (Weeks 1 to 18).
Time Frame: Week 1 to Week 18, Double-blind: weeks 1 to 18; Baseline: weeks -8 to -1; Titration: weeks 1 to 2; AED taper/conversion: weeks 3 to 8; Monotherapy: weeks 9 to 18
Population: efficacy population (ESL 1200 mg) Double-blind: 60; Baseline: 60; Titration: 60; AED taper/conversion: 60; Monotherapy: 43 (ESL 1600 mg) Double-blind: 118; Baseline: 118; Titration: 118; AED taper/conversion: 114; Monotherapy: 93
Measure: Mean (Standard Deviation); unit: Number of seizures in 28 days
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Number analyzed (Participants) | 65 | 128
Number of seizures in 28 days
  SSF during double-blind period | 8.8 (12.89) | 6.9 (6.50)
  SSF during baseline | 8.7 (5.63) | 10.9 (7.70)
  SSF during titration period | 6.2 (7.77) | 6.4 (7.53)
  SSF during AED taper/conversion period | 8.7 (14.78) | 6.9 (6.90)
  SSF during monotherapy period | 13.2 (29.52) | 6.8 (7.65)

ADVERSE EVENTS:
Time Frame: 18 weeks double-blind treatment period
Arm/Group | Eslicarbazepine 1200 mg QD | Eslicarbazepine 1600 mg QD
Serious Adverse Events (participants affected / at risk) | 4/65 | 8/128
Other Adverse Events (participants affected / at risk) | 46/65 | 100/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eslicarbazepine 1200 mg QD (N=65) | Eslicarbazepine 1600 mg QD (N=128)
cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Accidnetal overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral cyst (Nervous system disorders) | 0 (0) | 1 (1)
complex partial seizers (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eslicarbazepine 1200 mg QD (N=65) | Eslicarbazepine 1600 mg QD (N=128)
Diplopia (Eye disorders) | 5 (5) | 6 (6)
Vision blurred (Eye disorders) | 6 (6) | 12 (15)
Abdominal discomfort (Gastrointestinal disorders) | 4 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 9 (12)
Nausea (Gastrointestinal disorders) | 7 (9) | 18 (28)
Toothache (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7) | 11 (14)
Fatigue (General disorders) | 13 (14) | 20 (25)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 4 (4)
Influenza (Infections and infestations) | 4 (4) | 5 (5)
Nasopharyngitis (Infections and infestations) | 7 (7) | 14 (15)
Confusion (Injury, poisoning and procedural complications) | 4 (4) | 7 (8)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Dizziness (Nervous system disorders) | 18 (31) | 31 (42)
Headache (Nervous system disorders) | 14 (28) | 26 (33)
Memory impariment (Nervous system disorders) | 5 (5) | 2 (2)
Partial seizures with secondary generalisation (Nervous system disorders) | 6 (6) | 1 (1)
Somnolence (Nervous system disorders) | 7 (8) | 23 (33)
Insomnia (Psychiatric disorders) | 3 (3) | 8 (9)

LIMITATIONS AND CAVEATS:
The comparison of active treatment to control which was used in this trial is based on a pooled analysis of comparator groups from 8 earlier trials of similar design. Limitations related to use of historical control groups are applicable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish